CLINICAL TRIAL: NCT00718757
Title: A Phase I Trial Using Irinotecan, Vincristine, and Dexamethasone In Children With Relapsed And/Or Refractory Hematologic Malignancies
Brief Title: Irinotecan, Vincristine, and Dexamethasone In Children With Relapsed And/Or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIDML
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Non-Hodgkins Lymphoma; Hodgkin's Disease; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; Irinotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dexamethasone; Drug: Irinotecan; Drug: Vincristine

INTERVENTIONS:
Drug: Dexamethasone — 5 doses given on Days 6-10
Drug: Irinotecan — 20 mg/m2/day IV, 10 doses given on Days 1-5, 8-12
Drug: Vincristine — 1.5 mg/m2/day IV (max 2 mg), 2 doses given on Days 1,8
  * Patients < 1 year of age or < 10kg in weight: Vincristine 0.05 mg/kg

SUMMARY:
The purpose of this study is to estimate the maximum tolerated dose of dexamethasone given for 5 consecutive days when combined with fixed doses of irinotecan (given IV, qd x 5, 2 days off, qd x 5) and vincristine (given IV, 2 doses total on days 1 and 8 of schedule) in children with relapsed or refractory hematologic malignancies. In addition we will also study the pharmacokinetics of irinotecan when given without and then with dexamethasone in each patient, evaluate the relationship between irinotecan pharmacokinetic parameters and toxicity and describe any antitumor effects.

DETAILED DESCRIPTION:
TREATMENT PLAN

Treatment This is a phase I trial of irinotecan, vincristine, and dexamethasone administered over a 2-week period. Each treatment course will be a minimum of 21 days from the first day of irinotecan. Cycles may be repeated after hematologic recovery every 21 days if in the opinion of the primary physician the patient received some benefit from the chemotherapy. Irinotecan pharmacokinetic studies for each patient will be performed with the first course of therapy. From 4 to 18 patients will be treated to determine the MTD, irinotecan pharmacokinetics, and biologic effects of this combination of chemotherapeutic agents.

Drug Dosages for Each Course Irinotecan, 20 mg/m2/day IV, Days 1-5, 8-12

**Dexamethasone Days 6-10 Vincristine 1.5 mg/m2/day IV (max 2 mg), Days 1, 8 (patients < 1 year of age or < 10kg in weight: Vincristine 0.05 mg/kg)

CNS Chemotherapy

No intrathecal therapy will be given during the first course for any patients. Triple intrathecal chemotherapy (MHA) will be given on day 1 of subsequent courses (if patient is eligible) for patients with NHL or ALL. The age adjusted dosages are as follows:

<12 months Methotrexate 6 mg, Hydrocortisone 12 mg, Ara-C 18 mg 12 -24 months Methotrexate 8 mg, Hydrocortisone 16 mg, Ara-C 24 24-35 months Methotrexate 10 mg, Hydrocortisone 20 mg, Ara-C 30 ≥36 months Methotrexate 12 mg, Hydrocortisone 24 mg, Ara-C 36

**Dose Escalation for Dexamethasone

The doses for irinotecan and vincristine are fixed. The starting dose for dexamethasone will be 10 mg/m2/day po divided TID for 5 days. Intra-patient dose escalation will not be allowed.

Dose Level Dose (mg/m2/day) Dose Level 1 10 Dose Level 2 20 Dose Level 3 30 If the MTD is exceeded at the first dose level, then the subsequent cohort of patients will be treated at a dose that is 50% (5 mg/m2) lower than the starting dose.

Inter-Patient Escalation

Escalations are planned in groups of three patients, with up to three additional patients to be added at the first indication of DLT.

When 3 patients who are evaluable for toxicity have completed 3 weeks of therapy at a dose level without evidence of dose-limiting toxicity (DLT) subsequent patients may be enrolled at the next dose level.

If a dose-limiting toxicity is observed in 1 patient from the initial cohort of 3 patients at a given dose level, up to 3 additional patients will be entered at that dose level. If none of these additional patients experience a DLT (1/6 with DLT), the dose level will be escalated.

At the time a second patient has a DLT at a dose level (≥ 2 out of 2 to 6 patients), the MTD has been exceeded and the next lower dose will be considered the MTD.

If the MTD is exceeded at the first dose level, then the subsequent cohort of patients will be treated at a dose that is 50% (5 mg/m2) lower than the starting dose. If the MTD is exceeded at this lower level then the protocol will be stopped.

If the MTD is not reached, the maximum dose level studied will be considered the recommended dose.

The exception to the above escalation is if the dose-limiting toxicity is diarrhea in both patients required to define a MTD, then another cohort of patients will be treated at the same dose level with the addition of oral cefixime. If there are no dose-limiting toxicities in the cohort that receives cefixime, then dose escalation will continue as above with all further patients receiving oral cefixime.

Additional Courses

Patients may receive additional courses if in the opinion of the primary physician the patient received some benefit from the chemotherapy at intervals of 21 days as soon as hematologic recovery from the therapy has occurred. In addition, patients may receive intrathecal therapy as directed by the primary physician during these subsequent courses. Intra-patient escalation will not be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Age < or equal to 21 years at time of study entry
* Pathological diagnosis of a recurrent or refractory Non-Hodgkin's lymphoma, Hodgkin's disease, or acute lymphoblastic leukemia
* ECOG performance status < or equal to 2 (or Lansky play-performance scale > or equal to 50% for children <10 years of age).
* Has not received chemotherapy in previous 2 weeks. In the case of rapidly progressing disease, this criterion may be waived by consulting with the Principal Investigator, provided the patient has recovered from the acute effects of prior therapy.
* Hemoglobin >8 g/dl, absolute neutrophil count >1000 /mm3 (without growth factor support), and platelet count >50,000/mm3 (without transfusion support) unless bone marrow is involved with tumor or leukemia
* Adequate liver function (bilirubin < 1.5 x normal for age, AST and ALT < 3 x normal for age)
* Adequate renal function (serum creatinine <3 x normal for age)
* No active graft-versus-host disease (GVHD) or ongoing treatment for GVHD

Exclusion Criteria:

* Currently receiving other cytotoxic or investigational drugs
* Pregnant or lactating females are not eligible. Pregnancy tests must be obtained in females who are post-menarchal.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, azole antifungals, aprepitant, or St. John's Wort is not allowed.
* Evidence of active infection at the time of protocol entry
* History of allergy to any of the study medications

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose of dexamethasone given for 5 consecutive days when combined with fixed doses of irinotecan and vincristine in children with relapsed hematologic malignancies | Maximum Tolerated Dose (MTD)

CONTACTS AND LOCATIONS:
Overall Officials: John T Sandlund, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Rady's Children Hospital San Diego, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org